CLINICAL TRIAL: NCT03986008
Title: Effects of Benaglutide on Weight and Gut Microbiota in Obese Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019050125
Record Dates: First submitted 2019-06-11; First posted 2019-06-14 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Benaglutide (Experimental): Benaglutide will be administered three times a day by subcutaneous injection (under the skin) in the abdomen, thigh, or upper arm. It will be given 10 minutes before each meal.
  Interventions: Drug: Benaglutide
- Liraglutide (Active Comparator): Liraglutide will be administered once a day by subcutaneous injection (under the skin) in the abdomen, thigh, or upper arm. It will be given independently of meals and preferably at the same each day.
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Benaglutide — The treatment of Benaglutide lasted three months.During the first week: 0.1mg per day;During the second week: 0.14mg per day; From third week onwards, 0.2mg per day.
  Other Names: rhGLP-1(7-36)
  Arms: Benaglutide
Drug: Liraglutide — The treatment of Liraglutide lasted three months.During the first week: 0.6mg per day;During the second week: 1.2mg per day; From third week onwards, 1.8mg per day.
  Other Names: Victoza
  Arms: Liraglutide

SUMMARY:
The purpose of this studay is to evaluate the effects of Benaglutide on the treatment of subjects with obesity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 65 years (to the date of screening)；
2. The newly diagnosed obese patients (BMI greater than 28 kg/m2) or abdominal obesity (male waist circumference is greater than 90cm, female waist is greater than 85cm).
3. Nearly a month have not used weight-related drugs,including various weight-loss drugs,GLP-1 analogs or agonists,metformin, acarbose,insulin,anti hyperthyroid drugs,etc;Or recently used weight-related drugs but the stable dose was more than 1 month,and the drug dose remained constant or decreased during the trial.
4. Weight stable for more than 3 months (weight fluctuations <5%).

Exclusion Criteria:

1. pregnant female.
2. Secondary diseases caused by other diseases: including hypothyroidism, increased cortisol, hypothalamic and pituitary lesions caused by obesity, all kinds of drug-induced obesity, and others.
3. Severe cardiovascular and cerebrovascular diseases (heart failure, myocardial infarction, acute hemorrhagic or ischemic encephalopathy), pulmonary heart disease or pulmonary insufficiency, renal failure, severe hepatitis.
4. Combined with acute complications of diabetes such as ketoacidosis, lactic acidosis, hyperosmolar state of diabetes.
5. Nearly a month had surgery, trauma, infection and so on.
6. Limb deformity incomplete, difficult to accurately determine the height, weight and other physical indicators.
7. Poor medication compliance or serious side effects (severe rash, syncope, etc.).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-12-23 (Estimated); Study Completion 2021-12-23 (Estimated)

PRIMARY OUTCOMES:
Weight Change at 3 months | baseline and 3 months
  Measured in kilograms
Gut microbiota composition | 3 months
  Gut microbiota composition is assessed by 16S rRNA pyrosequencing. This analysis allows to obtain the relative abundance (%) of the different bacterial taxa and OTUs (operational taxonomic units).

SECONDARY OUTCOMES:
Change in waist circumference | baseline and 3 months
  Measured in cm
Change in systolic blood pressure | baseline and 3 months
  Measured in mmHg
Change in diastolic blood pressure | baseline and 3 months
  Measured in mmHg
Change in HbA1c | baseline and 3 months
  Measured in %
Change in plasma glucose | baseline and 3 months
  Measured in mmol/l
Change in insulin | baseline and 3 months
  Measured in μU/ml
Change in lipids-total cholesterol | baseline and 3 months
  Measured in mmol/l
Change in lipids-low density lipoprotein cholesterol | baseline and 3 months
  Measured in mmol/l
Change in lipids-high density lipoprotein cholesterol | baseline and 3 months
  Measured in mmol/l
Change in lipids-triglycerides | baseline and 3 months
  Measured in mmol/l
Change in lipids-free fatty acids | baseline and 3 months
  Measured in μmol/l
Change in Uric Acid | baseline and 3 months
  Measured in mmol/l
Change in interleukin-10 | baseline and 3 months
  Measured in mmol/l
Change in tumor necrosis factor | baseline and 3 months
  Measured in mmol/l

CONTACTS AND LOCATIONS:
Overall Officials: Jing Wu, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No